CLINICAL TRIAL: NCT04865705
Title: Neoadjuvant Chemotherapy and Tilelizumab in Stage III（cTNM-IIIA.IIIB）Non-small-cell Lung Cancer ,a Single-arm, Phase Ⅱ Clinical Trial
Brief Title: Neoadjuvant Chemotherapy and Tilelizumab in Stage III（cTNM-IIIA.IIIB）Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qinghua, Professor of Surgical Oncology and Molecular Biology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2020
Record Dates: First submitted 2020-10-26; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Stage III; Non-small Cell Lung Cancer
Keywords: stage III; driver gene negative; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tilelizumab+Albumin Paclitaxel + Carboplatin/Cisplatin (Experimental): Tilelizumab 200mg d1 Albumin Paclitaxel 260mg/m2 d1 Carboplatin/Cisplatin 75mg/m2/AUC5 d1IV,Q3W *2cycles
  Interventions: Drug: tislelizumab

INTERVENTIONS:
Drug: tislelizumab — Tilelizumab 200mg d1 Q3W Albumin Paclitaxel 260mg/m2 d1 Carboplatin/Cisplatin 75mg/m2/AUC5 d1 every 3 weeks
  Other Names: Albumin Paclitaxel; Carboplatin/Cisplatin

SUMMARY:
This is a prospective, one-arm, phase II study aimed at evaluating tislelizumab combined with platinum-containing dual-drug chemotherapy as a neoadjuvant treatment, supplemented with tislelizumab after surgery in patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
The study included a screening period, a treatment period (including neoadjuvant treatment, surgery and postoperative adjuvant treatment), and a survival follow-up period.

Patients who meet the admission criteria will receive the following treatments according to disease stage (IIIA/IIIB) and histology (squamous or non-squamous) Tilelizumab + platinum-containing dual-agent chemotherapy, every 3 weeks as a cycle , for 2 cycles, followed by surgical resection, and postoperative adjuvant Tilelizumab + platinum-containing dual-agent chemotherapy 2cycles,every 3 weeks as a cycle, and Tilelizumab every 3 weeks up to 15cycles maintenance treatment.

The rate of radical resection (R0) was evaluated through the research center of the investigator, which is expected to be 20% higher compared with historical controls, and the effectiveness of tislelizumab combined with platinum-containing dual-drug chemotherapy as a neoadjuvant treatment was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated and histologically confirmed stage III (T2N2, T3-4N1-2) NSCLC (as defined by the American Joint Committee on Cancer 8th Edition)
2. If the driver gene negative for EGFR sensitive mutations and ALK and ROS1 gene fusion mutations has not been detected before, test specimen tissue/blood
3. Tumor assessment scan using (CT) and (PET-CT) or magnetic resonance (MRI)
4. The date of signing the informed consent is ≥18 years old and ≤65 years old
5. Eastern Cooperative Oncology Group (ECOG) physical status is 0 or 1
6. Have measurable diseases assessed by the investigator according to RECIST Version 1.1
7. After neoadjuvant treatment, the MDT team and the chief surgeon comprehensively assessed and confirmed that they meet the requirements for radical resection
8. After neoadjuvant therapy, evaluate once every 2 cycles. For PD, discontinue tislelizumab and receive simultaneous radiotherapy. PR/SD patients will discuss MDT and adopt surgical treatment;
9. Good cardiopulmonary function, able to tolerate surgery
10. Eligible to receive platinum-containing dual-drug chemotherapy
11. Can provide representative pre-treatment tumor tissue samples/peripheral blood samples for biomarker analysis.

Exclusion Criteria:

1. Have received any treatment for the current lung cancer, including chemotherapy or radiotherapy 1.Patients with positive driver genes are known to carry EGFR mutations or ALK, ROS1 gene translocations
2. After neoadjuvant treatment, pneumonectomy is still required at the last evaluation
3. Suffered from any disease requiring systemic treatment with corticosteroids (daily dose of prednisone or equivalent drugs> 10 mg) or other immunosuppressive drugs in the 14 days before enrollment
4. Adrenaline replacement steroids (daily doses> 10 mg of prednisone or equivalent) are allowed for topical, ocular, intra-articular, intranasal or inhaled corticosteroids, and minimum systemic absorption is required, and they are prescribed Corticosteroids are short-term (≤7 days) medication, or used to treat non-autoimmune diseases
5. A history of active autoimmune disease or autoimmune disease that may recur.
6. Allow entry for patients with: well-controlled type I diabetes, hypothyroidism that requires only hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss), or predicted without external causes A disease that does not recur. The chest CT scan performed during the screening period has evidence of idiopathic pulmonary fibrosis, organic pneumonia (such as bronchiolitis obliterans), or a history of non-infectious pneumonia
7. Severe infections occurred within 4 weeks before enrollment, including but not limited to hospitalization due to infection complications, bacteremia or severe pneumonia
8. Severe chronic or active infections (including tuberculosis infection, etc.) that require systemic (oral or intravenous) antibiotic treatment within 14 days before enrollment
9. A history of interstitial lung disease, non-infectious pneumonia or poorly controlled diseases, including pulmonary fibrosis, acute lung disease, etc.
10. Untreated patients with chronic hepatitis B or HBV carriers with hepatitis B virus (HBV) DNA ≥ 500 IU/mL, or patients with active hepatitis C virus (HCV) should be excluded. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B carriers (HBV DNA <500 IU/mL), and cured hepatitis C patients can be included in the group.
11. If any major surgery requiring general anesthesia has been performed ≤28 days before randomization.
12. Previous allogeneic stem cell transplantation or organ transplantation. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Rate of radical resection (R0) | 2 weeks after neoadvant
  In the intention-to-treat (ITT) analysis set, the rate of radical resection (R0) is evaluated by the investigator, which is the number of people who can undergo R0 resection after the evaluation criteria established by the MDT team divided by the total number of enrolled groups

SECONDARY OUTCOMES:
PFS | up to 24-month
  The investigator evaluated the 24-month PFS to evaluate tislelizumab combined with platinum-containing dual-drug chemotherapy as a neoadjuvant treatment, and tislelizumab was added as an adjuvant treatment

OTHER OUTCOMES:
Biomarker level of PD-L1 | 2 weeks after surgery
  A PDL1 test measures the amount of PDL1 protein on cancer cells
Biomarker count of CD8+T cell | 2 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: yongseng wang, Principal Investigator — West China Hospital; qinghua zhou, Principal Investigator — West China Hospital
Locations (1):
- University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided